CLINICAL TRIAL: NCT07189884
Title: A Single-arm, Exploratory Clinical Study of Pyrotinib in Combination With Darcilib and Standard Endocrine Neoadjuvant Therapy for the Treatment of HR+HER2 Low-expression Breast Cancer
Brief Title: Pyrotinib Maleate Tablets in Combination With Dalpiciclib Isethionate Tablets and Standard Endocrine Therapy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-Ⅱ-246
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Breast Cancer (LABC)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib Maleate Tablets + Dalpiciclib Isethionate Tablets + Standard Endocrine (Experimental): Pyrotinib Maleate Tablets: 320 mg/day administered continuously from the first day of the first course of treatment, orally within 30 minutes after breakfast, missed doses without refill, every 21 days as a cycle.
  Dalpiciclib Isethionate Tablets: 125 mg orally every 28 days as a treatment cycle, with continuous medication for the first 3 weeks (Day 1 to Day 21), and rest (no medication) for the next 1 week (Day 22 to Day 28).
  Endocrine therapy: The endocrine therapy drug is selected by the investigator.
  Interventions: Drug: Pyrotinib Maleate Tablets + Dalpiciclib Isethionate Tablets + Standard Endocrine

INTERVENTIONS:
Drug: Pyrotinib Maleate Tablets + Dalpiciclib Isethionate Tablets + Standard Endocrine — Pyrotinib Maleate Tablets: 320 mg/day administered continuously from the first day of the first course of treatment, orally within 30 minutes after breakfast, missed doses without refill, every 21 days as a cycle.
  Dalpiciclib Isethionate Tablets: 125 mg orally every 28 days as a treatment cycle, with continuous medication for the first 3 weeks (Day 1 to Day 21), and rest (no medication) for the next 1 week (Day 22 to Day 28).
  Endocrine therapy: The endocrine therapy drug is selected by the investigator.

SUMMARY:
This study is a prospective, exploratory clinical study design, and plans to enroll 33 patients with HR+HER2 low expression breast cancer who received pyrotinib combined with darcili and standard endocrine neoadjuvant therapy to evaluate the efficacy of this regimen in HR+HER2 low expression breast cancer. Imaging evaluation was performed according to RECIST 1.1 criteria, and tumor imaging evaluation was performed by the participating center. The pathological evaluation after surgery of neoadjuvant patients was the pCR assessed by the pathologist of the participating center.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 years and ≤75 years old, who have just been treated for breast cancer;
2. Pathological examination confirmed that HR was positive (ER≥10%) and HER2 was low (immunohistochemical staining ICH++ and FISH negative);
3. Patients with invasive breast cancer confirmed by pathological examination (T≥3 or N≥1) who are eligible for neoadjuvant therapy;
4. ECOG score 0~1 points;
5. Planned to undergo definitive surgical resection of breast cancer, i.e., breast-conserving surgery or total mastectomy, sentinel lymph node (SN) biopsy, or axillary lymph node dissection (ALND);
6. Normal function of major organs, i.e. meeting the following criteria:

(1) Blood routine examination standards must meet: ANC ≥1.5×109/L; PLT ≥90×109/L； Hb ≥90g/L； (2) Biochemical examination must meet the following criteria: TBIL ≤upper limit of normal (ULN); ALT and AST ≤ 1.5 times the upper limit of normal (ULN), alkaline phosphatase ≤ 2.5 times the upper limit of normal (ULN), BUN and Cr ≤ 1.5× ULN and creatinine clearance ≥ 50 mL/min (CockcroftGault formula); (3) Cardiac color ultrasound and echocardiography: left ventricular ejection fraction (LVEF≥55%); (4) 18-lead ECG corrected by Fridericia's QT interval (QTcF) in women< 470 ms; 7. For female patients who are not menopausal or surgically sterilized: agree to abstain from sexual activity or use an effective contraceptive method during the treatment period and for at least 7 months after the last dose of study treatment; 8. Volunteer to join this study and sign the informed consent form.

Exclusion Criteria:

1. Those who have a known history of allergy to the drug components of this regimen;
2. Previous anti-tumor therapy or radiotherapy for any malignant tumor (except for cured cervical carcinoma in situ and basal cell carcinoma);
3. Underwent major surgical procedures unrelated to breast cancer within 4 weeks, or patients have not fully recovered from such surgical procedures;
4. Patients with stage IV (metastatic) breast cancer;
5. Inability to swallow, intestinal obstruction, or other factors affecting drug intake and absorption;
6. Severe heart disease or discomfort that cannot be treated;
7. Suffering from mental illness or psychotropic substance abuse and unable to cooperate;
8. Pregnant or lactating female patients;
9. Patients with severe liver and kidney function diseases and hematological diseases;
10. Those who are not suitable for enrollment in the investigator's opinion: such as a history of drug abuse, blood products, anticoagulant drugs and immunological drugs in the past year; Those with poor compliance and refusal to cooperate with treatment; Doctors with severe hypertension and diabetes are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-09-23 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 month
  Objective remission rate

IPD SHARING:
Plan to Share IPD: No